CLINICAL TRIAL: NCT05234723
Title: Epidemiological Burden of and Risk Factors for Ganciclovir Resistant Cytomegalovirus in Solid Organ Transplant Patients: Multicentre Cohort Study
Brief Title: Ganciclovir Resistant Cytomegalovirus Infection in SOT Recipients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ReCySOT
Record Dates: First submitted 2022-01-09; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Cytomegalovirus Infections
Keywords: Ganciclovir-resistant CMV; Cytomegalovirus; Solid Organ Transplant; Ganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ReCySOT study is a multicenter, retrospective, observational case-control study on risk factors for developing a ganciclovir-resistant (GCV-R) cytomegalovirus infection in patients receiving solid organ transplant. Aims of the study are to investigate the incidence of and risk factors for GCV-R CMV infection in SOT recipients in order to design further studies aimed at preventing and improving the patient management of GCV-R CMV infections.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is an important cause of morbidity and mortality in solid organ transplant (SOT) patients. Ganciclovir is the first line therapy for treatment and prevention of CMV infection in SOT recipients, with established efficacy and relatively safe profile.

Ganciclovir-resistant (GCV-R) CMV is an uncommon but frightening clinical problem due to limited, toxic and less effective therapeutic alternative drugs. Indeed, some studies indicate that GCV-R is associated with significant additional attributable morbidity and mortality in SOT recipients compared with ganciclovir susceptible (GCV-S) CMV disease.

Few data are available about the incidence of GCV-R-CMV in SOT patients showing a range from 0% to 3% . The serological mismatch group and the type of SOT have been reported as the main factors influencing such range. Indeed, in one of the largest experience now available, the incidence of GCV-R accounted up to 12% in a cohort of lung transplant recipients.Risk factors for ganciclovir resistance development appear to be the high-risk D+/R- subset, high viral loads, increased durations of antiviral drug exposure and the use of more potent immunosuppression. However, these reports come from small, monocentric experiences with a limited number of cases.

In general, mutations that confer resistance to ganciclovir are not present at baseline but emerge and become amplified over time, especially in the presence of an incompletely suppressive drug exposure. The GCV-R is due to mutations in UL97 and UL54 genes. UL97 mutations confer various degrees of phenotypic resistance to ganciclovir. Mutations in UL54 determine higher-level resistance to ganciclovir and usually appear as a second step after mutations in UL97.

Second-line strategies for the treatment of GCV-R CMV are based on high dose of GCV administration or foscarnet/cidofovir use, both with a high risk of metabolic and renal dysfunction. Alternative strategies are based on the use of adjunctive treatments such as cytomegalovirus immunoglobulins (IVIG), infusions of CMV-specific Tcells or several drugs with indirect anti-CMV action (mTOR inhibitors sirolimus and everolimus, leflunomide and artesunate). Finally, the new antiviral drugs approved for prophylaxis (letermovir) or in advanced clinical development (maribavir, brincidofovir), are reported as anecdotical alternative strategies for the treatment of GCV-R CVM infection. The limited therapeutic strategies for GCV-R CMV treatment highlight the need for new strategies to prevent resistance development.

The investigators carry-out a multicenter retrospective observational study to define incidence of GCV-R CMV-infection in SOT patients and to identify the risk factors for its development in SOT recipients. Data from this study could be useful to design further studies aimed at preventing and improving the patient management of GCV-R CMV infections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CMV infection in adult (age ≥ 18 years) patients underwent SOT
* Ability to understand the purpose of the study and provide signed and dated informed consent

Exclusion Criteria:

* Lack of clinical and/or laboratory data to establish the type of CMV event
* Lack of the serological mismatch at transplantation
* Lack of the type of SOT
* Lack of the patient and graft outcome at 30, 60 or 90 days after CMV event diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥ 18 years) patients who underwent SOT developing CMV-infection during the study period will be screened for inclusion according to inclusion and exclusion criteria. Eligible patients will be classified as cases or controls according to the following definitions:
  * Case: SOT recipients with genotypically confirmed GCV-R CMV-event;
  * Control: SOT recipients with "presumed" GCV-S CMV-event on the basis of good microbiological and clinical response to standard GCV/VGC treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
To define incidence of GCV-R CMV-infection in SOT patients | Through study completion, an average of 1 year
  To define incidence of GCV-R CMV-infection in SOT patients
To define the risk factors for GCV-R CMV-infection development in SOT patients | Through study completion, an average of 1 year
  To define the risk factors for GCV-R CMV-infection development in SOT patients

SECONDARY OUTCOMES:
To compare type of CMV episode between SOT patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To compare type of CMV episode: infection or disease (the last cathegorized as CMV syndrome or Tissue invasion) between SOT patients with GCV-R versus GCV-S CMV-infection.
To compare virological cure between SOT patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To compare virological cure at 30, 60 and 90 days after CMV infection diagnosis and relapse of CMV infection between SOT patients with GCV-R versus GCV-S CMV-infection.
To compare clinical cure between SOT patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To compare clinical cure at 30, 60 and 90 days after CMV infection diagnosis between SOT patients with GCV-R versus GCV-S CMV-infection.
To compare graft outcome between SOT patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To compare graft failure rate and the need of re-SOT between SOT patients with GCV-R versus GCV-S CMV-infection between SOT patients with GCV-R versus GCV-S CMV-infection.
To compare the need of ICU and hospital stay between SOT patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To compare total length of ICU and hospital stay between SOT patients with GCV-R versus GCV-S CMV-infection.
To compare the need of readmission in ICU and/or hospital between SOT patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To compare the need of readmission in ICU and/or hospital between SOT patients with GCV-R versus GCV-S CMV-infection.
To compare all cause mortality between SOT patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To compare all-cause mortality during infection episode and follow-up (30, 60, 90 days after the first CMV infection diagnosis) between SOT patients with GCV-R versus GCV-S CMV-infection.
To describe the therapeutic management of GCV-R CMV-infection. | Through study completion, an average of 1 year
  To describe the therapeutic management of GCV-R CMV-infection.
To evaluate differences of CMV-specific T-cell response in patients with GCV-R versus GCV-S CMV-infection. | Through study completion, an average of 1 year
  To evaluate differences of CMV-specific T-cell response in patients with GCV-R versus GCV-S CMV-infection. CMV-specific T-cell response will be assesed determining the detection of IFN-γ expressed in UI/ml after stimulation of whole blood or peripheral blood mononuclear cells (PBMC) with CMV-specific antigens or overlapping peptides.